CLINICAL TRIAL: NCT04118985
Title: Compensatory Training to Support Everyday Function and Adherence to Brain Healthy Lifestyle Changes in Those at Risk for Alzheimer's Disease
Brief Title: Compensatory Training to Support Brain Healthy Lifestyle Changes in Those at Risk for Alzheimer's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Dona E. Locke, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 19-006676
Record Dates: First submitted 2019-09-08; First posted 2019-10-08 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Cognitive Symptom; Pre Senile Dementia; Alzheimer Disease
Keywords: Subjective cognitive complaint
MeSH Terms: conditions — Neurobehavioral Manifestations; Alzheimer Disease | interventions — Cognitive Training

STUDY DESIGN:
Intervention Model Description: Randomized to one of 1 arms: 1) provided recommendations and materials without coaching for implementation 2) provided recommendations and materials with 10 coaching classes
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-implementation (Active Comparator): Individuals randomized to this group will be given all the materials about cognitive compensations techniques and brain health behavior guidelines and encouraged to implement those on their own.
  Interventions: Behavioral: Self-implementation
- Health-behavior intervention (Experimental): Individuals randomized to this group will attend 10 weekly classes designed to provide information about cognitive compensation techniques and brain health behaviors as well as interventional support to implement those recommendations with homework and follow-up classes.
  Interventions: Behavioral: Cognitive rehabilitation and health behavior change intervention

INTERVENTIONS:
Behavioral: Cognitive rehabilitation and health behavior change intervention — Cognitive rehabilitation and health behavior change intervention in a group-based program intervention compared to self-implementation of techniques without these interventions
  Arms: Health-behavior intervention
Behavioral: Self-implementation — Self-implementation of cognitive rehabilitation and health behavior change recommendations
  Arms: Self-implementation

SUMMARY:
The Researchers are trying to better understand if behavioral interventions can help improve memory compensation and engagement in healthy lifestyle behaviors in those with memory concerns but normal mental status exam.

ELIGIBILITY:
Inclusion Criteria:

* Age 50 or older
* A positive complaint or concern in response to two questions ('Do you feel like your memory or other aspects of thinking are becoming worse?' and 'Does this worry you?')
* Normal cognitive performance on the Montreal Cognitive Assessment (adjusted for age and education)
* Self-reported independent function in daily life as measure by the Lawson IADL scale (IADL=8)
* English speaking
* Approval letter from a physician (due to the exercise component)

Exclusion Criteria:

* Known neurological disorder with potential cognitive symptoms (a diagnosis of Parkinson's disease, epilepsy, a history of significant TBI, etc.)
* Uncontrolled moderate or severe depression (e.g., CES-D > 21).

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-10-10 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Everyday Compensation Questionnaire | baseline, change from baseline at end of 10 week treatment, change from baseline at 3 months, change from baseline at 6 months
  self-report and informant report if an informant is available of compensatory strategy use; range 0-148 with higher scores indicating more compensatory use
Lifestyle Activities Questionnaire | baseline, change from baseline at end of 10 week treatment, change from baseline at 3 months, change from baseline at 6 months
  self-report of cognitive activities, range 13-65 with higher scores indicating more activity
BrainHQ | baseline, change from baseline at end of 10 week treatment, change from baseline at 3 months, change from baseline at 6 months
  Number of minutes on BrainHQ computer exercise program
Physical Activities Questionnaire | baseline, change from baseline at end of 10 week treatment, change from baseline at 3 months, change from baseline at 6 months
  self-report of physical activity; scores include number of days per week across 7 activity types and number of minutes in each activity when completed.
Mindful Attention Awareness Scale | baseline, change from baseline at end of 10 week treatment, change from baseline at 3 months, change from baseline at 6 months
  self-report of mindfulness, range of 11-66 with higher scores indicating more mindful daily experience

SECONDARY OUTCOMES:
Everyday Cognition | baseline, change from baseline at end of 10 week treatment, change from baseline at 3 months, change from baseline at 6 months
  self-report of everyday functioning, range 39-156 with higher scores indicating more problems in daily functioning
Quality of Life (in aging and cognitive health) | baseline, change from baseline at end of 10 week treatment, change from baseline at 3 months, change from baseline at 6 months
  self-report of quality of life, range of 13-52 with higher scores indicating better quality of life
Psychological well-being | baseline, change from baseline at end of 10 week treatment, change from baseline at 3 months, change from baseline at 6 months
  self-report of psychological well-being/happiness; there is a total score plus subscales of autonomy, environmental mastery, personal growth, positive relations with others, purpose in life, self-acceptance. Each subscale has 9 items for a total of 54 items. Total scores range from 54-324 with higher scores indicating higher psychological well being. Each subscale ranges from 9-54 with higher scores indicating greater well-being on that construct.
Centers for Epidemiological Studies - Depression | baseline, change from baseline at end of 10 week treatment, change from baseline at 3 months, change from baseline at 6 months
  self-report of symptoms of depression.Range 0-60 with higher scores indicating more depression
Cognitive measure of memory | baseline, change from baseline at end of 10 week treatment, change from baseline at 3 months, change from baseline at 6 months
  Hopkins Verbal Memory test. Staff administered standardized verbal memory task. Scores include total words recalled and total recalled after a delay with higher scores indicating greater recall
cognitive measure of executive functioning | baseline, change from baseline at end of 10 week treatment, change from baseline at 3 months, change from baseline at 6 months
  Trailmaking test; Staff administered standardized measure of attention and executive functioning. Scores include time to complete the task (with higher scores being slower) and number of errors
cognitive measure of verbal fluency | baseline, change from baseline at end of 10 week treatment, change from baseline at 3 months, change from baseline at 6 months
  Controlled Oral Word Association Test; Staff administered standardized measure of speed and verbal fluency. Score is number of items in one minute with higher scores indicating better functioning
cognitive measure of visual scanning speed | baseline, change from baseline at end of 10 week treatment, change from baseline at 3 months, change from baseline at 6 months
  Symbol Digit Modalities Test; Staff administered standardize measure of speed and visual scanning. Scores indicate number of items completed in the time frame with higher scores indicating better functioning.
cognitive measure of response inhibition | baseline, change from baseline at end of 10 week treatment, change from baseline at 3 months, change from baseline at 6 months
  Stroop Color Word Test; Staff administered standardized measure of speed and response inhibition. Scores indicate number of items completed in the time limit with higher scores indicating better functioning

CONTACTS AND LOCATIONS:
Overall Officials: Dona Locke, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Scottsdale, Arizona, United States

IPD SHARING:
Plan to Share IPD: No
The study is quite small and is meant a pilot data for preliminary feasibility and effect size estimating.

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-22): https://cdn.clinicaltrials.gov/large-docs/85/NCT04118985/Prot_SAP_000.pdf